CLINICAL TRIAL: NCT00053144
Title: Irinotecan And Cytarabine In Refractory or Relapsed Acute Myeloid Leukemia And In Chronic Myelogenous Leukemia In Myeloid Blast Transformation: Efficacy And In Vitro Correlates
Brief Title: Irinotecan and Cytarabine in Treating Patients With Refractory or Recurrent Acute Myeloid Leukemia or Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Maria Baer, Roswell Park Cancer Institute
Purpose: Treatment
Other Study IDs: CDR0000269286; P30CA016056 (NIH); RPCI-RPC-9901
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; Philadelphia chromosome positive chronic myelogenous leukemia; secondary acute myeloid leukemia; blastic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; adult acute monocytic leukemia (M5b); adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute promyelocytic leukemia (M3)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute | interventions — Cytarabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cytarabine
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of combining irinotecan with cytarabine in treating patients who have refractory or recurrent acute myeloid leukemia or chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity of irinotecan and cytarabine in patients with refractory or recurrent acute myeloid leukemia or chronic myelogenous leukemia in myeloid blast transformation.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine the maximum tolerated dose of irinotecan in this regimen in these patients.
* Correlate the clinical activity of this drug with cellular endpoints associated with DNA synthesis inhibition, DNA repair, induction of apoptosis, and drug resistance in these patients.

OUTLINE: This is a dose-escalation study of irinotecan.

Patients receive irinotecan IV over 90 minutes and cytarabine IV over 60 minutes on days 1-6. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. An additional 9 patients with refractory/relapsed acute myeloid leukemia and 9 patients with chronic myelogenous leukemia in myeloid blast transformation are treated at the MTD.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 3-36 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute myeloid leukemia (M0-M7)

  * De novo or secondary disease

    * Previously treated and refractory to prior therapy (which has included high-dose cytarabine and an anthracycline)
  * Antecedent hematologic disorders allowed OR
* Histologically confirmed Philadelphia chromosome-positive chronic myelogenous leukemia in myeloid blast transformation

  * Treated or untreated
  * Blast transformation defined by at least 20% blasts in marrow and/or blood
  * Myeloid lineage defined by immunophenotyping

PATIENT CHARACTERISTICS:

Age

* 15 and over

Performance status

* 0-3

Life expectancy

* At least 4 weeks

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin less than 2 times upper limit of normal (ULN)
* SGOT less than 2 times ULN

Renal

* Creatinine less than 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* No other concurrent serious medical or psychiatric illness that would preclude study consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* Prior chemotherapy for an antecedent malignancy or other medical condition allowed

Endocrine therapy

* Not specified

Radiotherapy

* Prior radiotherapy for an antecedent malignancy or other medical condition allowed

Surgery

* Not specified

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-11; Primary Completion 2003-02 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria R. Baer, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States